CLINICAL TRIAL: NCT05068856
Title: A Phase I, Multi-Center, Open Label, Dose Escalation/Expansion Study of HRS2543 in Patients With Advanced Tumors
Brief Title: A Study of HRS2543 in Patients With Advanced Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: R&d strategy adjustment
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS2543-I-101
Record Dates: First submitted 2021-09-15; First posted 2021-10-06 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Advanced Tumors

STUDY DESIGN:
Intervention Model Description: HRS2543 monotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS2543 (Experimental)
  Interventions: Drug: HRS2543

INTERVENTIONS:
Drug: HRS2543 — Dose-escalation part For the dose-escalation study, five dose cohorts (25 mg , 75 mg , 150 mg , 300 mg , and 450 mg ) of HRS2543 are initially set.
  Dose-expansion part After the completion of dose-escalation study, the dose-expansion study will be carried out at the recommended dose level by the SMC.

SUMMARY:
To assess the safety and tolerability of HRS2543 in patients with advanced tumors and to determine the recommended phase II dose (RP2D) of HRS2543

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years of age, both male and female
2. non standard treatment, invalid the standard treatment or refuse to receive standard treatment in patients with advanced tumors diagnosed by pathology
3. the Eastern Cooperative Oncology Group （ECOG） General status (performance status, PS) of 0-1
4. the expected lifetime ≥ 3 months
5. Has at least one measurable lesion as defined by RECIST v1.1
6. Written informed consent is provided by signing the informed consent form

Exclusion Criteria:

1. Any previous anti-tumor treatment
2. The toxicity caused by any previous anti-tumor treatment has not recovered to ≤ grade 1
3. Any other anti-tumor treatment is planned during the study treatment
4. After imaging diagnosis, there were brain tumor lesions
5. According to the judgment of the researcher, there are factors that can not swallow, chronic diarrhea and intestinal obstruction or other factors that can significantly affect the absorption, distribution, metabolism or excretion of drugs
6. Active heart disease was present within 6 months before the first administration of the study
7. Other malignancies occurred within 5 years before the first administration of the study
8. Active HBV or HCV infection
9. The subject had a history of immune deficiency
10. According to the judgment of the researcher, there are concomitant diseases that seriously endanger the safety of the subjects, confuse the analysis of the test results, or affect the subjects to complete the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | Day 1 to 28 (Cycle 1)
  A DLT is considered at AE related to study drug unless there is a clear, well-documented, alternative explanation for the toxicity. Severity of AEs are graded according to the NCI CTCAE 5.0 for the study, the occurrence of the following drug related AEs during the single dose and the first cycle (28 days) will be considered a DLT by the investigator and SMC.
Maximum Tolerated Dose (MTD) | Day 1 to 28 (Cycle 1)
  Toxicity will be evaluated according to the NCI CTCAE Version 5.0.
Recommended PhaseII Dose (RP2D) | Day 1 to 28 (Cycle 1)
  Toxicity will be evaluated according to the NCI CTCAE Version 5.0.

SECONDARY OUTCOMES:
Number of patients with changes in laboratory measurements | up to 24 months
Number of patients with changes in single and triplicate 12-lead Electrocardiogram (ECG). | up to 24 months
Number of patients with changes in ECOG PS score. | up to 24 months
Number of patients with changes in Physical Examination. | up to 24 months
Number of patients with changes in Vital Signs | up to 24 months
Incidence of adverse events (AEs). | up to 24 months
Cmax of HRS2543 after single dose of HRS2543 | Day 1 of Cycle 1(each cycle 28 days)
Tmax of HRS2543 after single dose of HRS2543 | Day 1 of Cycle 1(each cycle 28 days)
AUC0-t of HRS2543 after single dose of HRS2543 | Day 1 of Cycle 1(each cycle 28 days)
AUC0-∞ of HRS2543 after single dose of HRS2543 | Day 1 of Cycle 1(each cycle 28 days)
t1/2 of HRS2543 after single dose of HRS2543 | Day 1 of Cycle 1(each cycle 28 days)
Vz/F of HRS2543 after single dose of HRS2543 | Day 1 of Cycle 1(each cycle 28 days)
CL/F of HRS2543 after single dose of HRS2543 | Day 1 of Cycle 1(each cycle 28 days)
Cmax,ss of HRS2543 after multiple dose administration of HRS2543 | Up to 4 cycles (each cycle 28 days)
Tmax,ss of HRS2543 after multiple dose administration of HRS2543 | Up to 4 cycles (each cycle 28 days)
Cmin,ss of HRS2543 after multiple dose administration of HRS2543 | Up to 4 cycles (each cycle 28 days)
AUCss of HRS2543 after multiple dose administration of HRS2543 | Up to 4 cycles (each cycle 28 days)
Rac of HRS2543 after multiple dose administration of HRS2543 | Up to 4 cycles (each cycle 28 days)
ORR: the Objective Response Rate | up to 24 months
DoR: the Duration of Response | up to 24 months
DCR: the Disease Control Rate | up to 24 months
PFS: the Progression Free Survival | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiao Tong University School of Medicine, Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided